CLINICAL TRIAL: NCT00236483
Title: A Comparison of the Efficacy and Safety of ULTRACET® (Tramadol HCl/Acetaminophen) Versus ULTRAM® (Tramadol HCl) Versus Placebo in Subjects With Pain Following Oral Surgery
Brief Title: A Comparison of the Effectiveness and Safety of ULTRACET® (Tramadol Hydrochloride/Acetaminophen) Versus ULTRAM® (Tramadol Hydrochloride) Versus Placebo in Patients With Pain After Oral Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002806
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Surgery, Oral; Pain, Postoperative
Keywords: Oral Surgery; Analgesics; Postoperative Pain; dental
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultracet

INTERVENTIONS:
Drug: tramadol hydrochloride + acetaminophen

SUMMARY:
The purpose of this study is to explore the pain-relieving effects and safety of two analgesic treatment regimens as compared to placebo in patients experiencing pain after oral surgery. Tramadol hydrochloride/acetaminophen is approved to treat acute pain. This study will evaluate the effectiveness and safety of tramadol hydrochloride/acetaminophen compared with tramadol hydrochloride alone compared with placebo as a pain medication in the treatment of pain following oral surgery.

DETAILED DESCRIPTION:
While other studies have shown the effectiveness and safety of tramadol/acetaminophen and of tramadol alone in treating pain following oral surgery, a direct comparison of the two treatments within the same study at these dose levels has not be performed. This is a single-center, randomized, double-blind, active- and placebo-controlled, single-dose, parallel-group study of adult patients who undergo oral surgery for removal of two or more impacted third molars. Patients who have at least moderate pain within 5 hours after surgery will be given a single oral dose of 2 capsules of study medication. Patients will be equally assigned to receive a total dose of either tramadol HCl 75 mg/acetaminophen 650 mg or tramadol HCl 100 mg or placebo. Patients will be asked about the intensity of the current pain and pain relief from the starting pain at 30 minutes and at 1, 2, 3, 4, 5 and 6 hours after taking the study medication. Patients will also be given two stopwatches that will be started once medication has been taken. Patients will stop the first stopwatch when they first notice any pain decrease; they will stop the second stopwatch when they notice meaningful pain relief. The primary efficacy endpoints are summary measures of hourly patient reported pain relief (PAR) and pain intensity scores: total PAR (TOTPAR), sum of hourly pain intensity differences (PIDs) from baseline (SPID), and sum of hourly PAR plus hourly PIDs from baseline (SPRID). The study hypothesis is that pain relief with tramadol HCl/acetaminophen (ULTRACET®) is superior to pain relief from tramadol HCl (ULTRAM®) alone after oral surgery and the combination is well tolerated.

2 capsules, total dose either tramadol HCl 75 milligrams/acetaminophen 650 milligrams, tramadol HCl 100 milligrams, or matching placebo taken one time orally; all study medication is over-capsulated to match.

ELIGIBILITY:
Inclusion Criteria:

* Surgical procedure involving removal of >= 2 impacted third molars with bone removal required for at least 2 of the 3 impacted third molars
* At least moderate pain within 5 hours after oral surgery procedure
* Sufficiently alert to follow directions, communicate with study personnel and perform study procedures
* If female, using an acceptable method of birth control and has a negative urine pregnancy test

Exclusion Criteria:

* Previously treated patients who have discontinued treatment due to an adverse event
* Patients who have had inadequate pain relief from tramadol HCl/acetaminophen or tramadol
* Patients who have used pain medication (other than anesthesia) within 24 hours of receiving study medication, any long-acting over-the-counter pain medications within 3 days, or any pain medication after finishing oral surgery
* Patients with known problems with taking opioid medications or acetaminophen
* Patients with a history of abusing drugs or alcohol
* Patients with an uncontrolled medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2002-11; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of total pain relief (TOTPAR), sum of pain intensity differences (PIDs) from baseline (SPID), and sum of total of pain relief and pain intensity differences (SPRID), 0 (baseline) to 6 hours after taking the study medication.

SECONDARY OUTCOMES:
Evaluations of hourly pain relief (PAR); duration of pain relief; times to onset of any noticable decrease in pain and meaningful pain relief, time to remedication; patient overall medication assessment; and safety evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Fricke JR Jr, Hewitt DJ, Jordan DM, Fisher A, Rosenthal NR. A double-blind placebo-controlled comparison of tramadol/acetaminophen and tramadol in patients with postoperative dental pain. Pain. 2004 Jun;109(3):250-257. doi: 10.1016/j.pain.2004.01.004. PMID 15157685
- See also: A COMPARISON OF THE EFFICACY AND SAFETY OF ULTRACET (TRAMADOL HCL/ACETAMINOPHEN) VERSUS ULTRAM® (TRAMADOL HCL) VERSUS PLACEBO IN SUBJECTS WITH PAIN FOLLOWING ORAL SURGERY — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=489&filename=CR002806_CSR.pdf